CLINICAL TRIAL: NCT06909903
Title: Cell Content of Sputum Induced by Hypertonic Saline in Adolescents With Cystic Fibrosis
Acronym: OCSI-CF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty including the last participants
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-60
Record Dates: First submitted 2025-03-11; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Within-subject crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Spontaneous sputum followed by sputum induced by Hypertonic Saline (Other): Part 1: At 9:00 a.m., we begin the physiotherapy session in the form of autogenic drainage for 30 minutes, then collection of secretions (ECBC No. 1 in two 40 mL CBC pots). The order of the physiotherapy sessions, with and without SSH, was decided based on the possible interactions between the two proposed treatments. SSH nebulization has a prolonged fluidifying effect over several hours and could influence the collection of secretions. Autogenic drainage would have the same effect, but for a maximum duration of 2 to 3 hours. The patient continues the usual course of visits to the CRCM.
  Part 2: At 2:00 p.m., we set up the protocol for expectoration induced by SSH nebulization, then we perform autogenous drainage for 30 minutes and collect the secretions (ECBC No. 2 in two 40 mL CBC pots). One of the pots is sent to Pr Roll's cytology laboratory and the other to Pr Drancourt's bacteriology laboratory within 30 minutes.
  Interventions: Procedure: Autogenous drainage of sputum caused by hypertonic saline in adolescents with cystic fibrosis.

INTERVENTIONS:
Procedure: Autogenous drainage of sputum caused by hypertonic saline in adolescents with cystic fibrosis. — The procedure will be performed at the same session as follows :
  * 30 minutes of autogenous drainage, followed by collection of secretions.
  * 10 minutes of HSS followed by 30 minutes of autogenous drainage before secretions are collected.
  The intervention first step involves verifying patient tolerance to Hypertonic saline solution nebulization (Auscultation, peak flow, saturtion levels), followed by the inhalation of 2 puffs of Ventolin® to prevent bronchospasm. Ten minutes later, the patient undergoes a 10-minute nebulization of 4 mL SSH 6% carried out according to the HAS recommendations.
  The patient tolerance to SSH is reassessed. If there are no adverse reactions, the patient continues the protocol. If issues like wheezing, a ≥5% drop in SpO2, or a ≥20% drop in Peak Flow occur, 4 more puffs of Ventolin® are given, and the patient is reassessed.If still intolerant, the patient exits the study.
  The session ends with physiotherapy (autogenous drainage) to aid mucus clearance.

SUMMARY:
Cystic fibrosis requires regular monitoring of bacterial colonization of sputum. The collection is done during scheduled consultations or urgently during exacerbations during the respiratory physiotherapy session, which is increasingly often associated with nebulization of Hypertonic Salt Serum (SSH). This allows, compared to simple expectoration, to obtain a greater density and diversity of germs. However, no study has focused on researching the precise place of origin of the collected secretions. Our aim is therefore to compare, in this pilot study in 20 adolescents suffering from cystic fibrosis and regularly followed at the pediatric CRCM, the ratio between squamous cells (CM, ENT origin) and broncho-alveolar cells in sputum obtained spontaneously and induced with of the SSH (collaboration with Professor Roll). The secondary criteria are the CM/bronchial cell ratio, the CM/alveolar macrophage ratio, cell viability and microbiological diversity. The hypothesis of this research is as follows: the nebulization of SSH before expectoration makes it possible to obtain a greater quantity of secretions from the broncho-alveolar sphere than during simple expectoration. In the cohort of 165 patients followed at the pediatric CRCM of Marseille, only 25 patients correspond to the inclusion criteria: they are between 12 and 17 years old, master autogenous drainage as well as spontaneous expectoration in sufficient quantity to carry out the research. They must also have been in stable clinical condition for at least one month. Taking into account the non-inclusion criteria (refusal to participate, systemic antibiotic therapy, respiratory decompensation or upper airway infection, SpO2 less than 92% before nebulization, appearance of hemoptysis in the last three months), the number of subjects is fixed. To 20. Each patient participates in a single day of hospitalization scheduled at the pediatric CRCM: at 9 a.m. simple expectoration and at 1 p.m., expectoration caused by SSH. The subject is therefore his own witness. The study inclusion period is one year.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent between 12 and 17 years old with definite cystic fibrosis (two CFTR gene mutations identified and positive sweat test)
* Patient followed at the pediatric CRCM of Marseille
* Patient able to expectorate spontaneously and master autogenous drainage
* Patient in stable clinical condition for 1 month

Exclusion Criteria:

* Patient refusing the study
* Patient under systemic antibiotic therapy
* Patient with respiratory decompensation or upper airway infection
* Patient with oxygen saturation < 92% before nebulization
* Patient with hemoptysis in the last 3 months
* Patients with decompensated heart failure

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 17 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-10-10 (Actual)

PRIMARY OUTCOMES:
Efficiency of 2 methods of secretion collection by assessing the percentage of squamous cells compared to the percentage of bronchoalveolar cells | Visit 0 at Month 0
  Compare, in adolescents with cystic fibrosis, the efficiency of 2 methods of secretion collection (during spontaneous sputum or during sputum induced by HSS) concerning the origin of the collected secretions judged by the study of the distribution of cells of the ENT sphere (squamous cells - SC) and of bronchoalveolar cells.

SECONDARY OUTCOMES:
Ratio of squamous cells to bronchial cells by cytological analysis of sputum samples | Visit 0 at Month 0
Ratio of squamous cells to alveolar macrophages by cytological analysis of sputum samples | Visit 0 at Month 0
Observe cell viability by assessing the percentage of dead cells | Visit 0 at Month 0
Assess the density and microbiological diversity of sputum | Visit 0 at Month 0

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hôpitaux de Marseille; Jean-Christophe DUBUS, Principal Investigator — CHU Timone Enfants
Locations (1):
- Médecine Physique et réadaptation - CHU Timone Enfants, Marseille, France, France

IPD SHARING:
Plan to Share IPD: No